CLINICAL TRIAL: NCT00646581
Title: Effect of Single Dose Intranasal Insulin on Cognitive Function in Patients With Schizophrenia
Brief Title: Effect of Single Dose Intranasal Insulin On Cognitive Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Xiaoduo Fan, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4-2006; CORRC tracking number: 4-2006
Record Dates: First submitted 2008-01-31; First posted 2008-03-28 (Estimated); Results first posted 2013-01-29 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Memory; Concentration; Insulin
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Insulin Resistance | interventions — Insulin; Insulin, Regular, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (1) (Placebo Comparator): Subjects are given a one-time, single dose of placebo intranasal spray
  Interventions: Drug: Placebo
- Single-Dose Intranasal Insulin (Experimental): Subjects are given a one-time, single dose of intranasal insulin
  Interventions: Drug: Insulin (Humulin)

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo (1)
Drug: Insulin (Humulin) — 40 IU Intranasal Insulin will be administered once
  Other Names: Humulin
  Arms: Single-Dose Intranasal Insulin

SUMMARY:
The purpose of the study is to find out how a small dose of insulin might affect memory, the ability to concentrate, and improve your daily functioning in patients with schizophrenia and schizoaffective disorders. Insulin is not being used to treat diabetes in this study. The investigators propose a single dose, double-blinded, placebo-controlled trial of intranasal insulin in 40 subjects with schizophrenia or schizoaffective disorder to examine insulin's effect on cognition. The specific aims include:

1. Examine the effects of single doses of 40 IU intranasal insulin compared to placebo on cognitive functioning, including attention and memory.
2. Examine whether single dose of intranasal insulin administration will raise serum insulin level and decrease plasma glucose level

Insulin will be delivered through an air spray pump into your nose. The investigators will be comparing one dose of insulin (40 International Units) with placebo, an inactive liquid.

DETAILED DESCRIPTION:
Insulin signaling in the brain is associated with improved cognitive function in both animal and human studies. Intranasal administration of insulin, which is non-invasive and minimizes the risk of hypoglycemia, may represent a new intervention approach with the potential to improve cognition and real life functioning in this patient with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Diagnosis of schizophrenia, any subtype or schizoaffective disorder, any subtype
* Male or female
* Stable dose of the current antipsychotic drug for at least one month
* Well established compliance with out-patient treatment per treating clinician's judgement.
* Able to complete the cognitive assessment battery (must be English speaking)

Exclusion Criteria:

* Inability to provide informed consent
* Current substance abuse
* On clozapine or olanzapine
* Psychiatrically unstable per treating clinician's judgement.
* Significant medical illnesses including uncontrolled hypertension, diabetes, seizure disorder, severe cardiovascular, cerebrovascular, pulmonary, or thyroid diseases etc.
* Incapable to complete the cognitive battery assessment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoduo Fan, MD, MPH, MS, Principal Investigator — UMass Medical School
Locations (1):
- Freedom Trail Clinic, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from an urban community mental health clinic.
Pre-assignment Details: Subjects who met DSM-IV criteria for schizophrenia or schizoaffective disorder were enrolled in the study (see inclusion/exclusion criteria). Subjects were randomly assigned to either the experimental group or placebo group.
Period: Overall Study
Arm/Group | Placebo (1) | Single-Dose Intranasal Insulin
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (1) | Single-Dose Intranasal Insulin | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Cognitive Function- HVLT Immediate Recall Total (Number)
Description: Subjects performed the HVLT Immediate Recall Task. For this task, participants were read aloud a list of 12 words from three taxonomic categories. Participants were read the list three separate times, and after each reading were immediately asked to recall as many words from the list as they could. The number of words recalled successfully was measured before and after intranasal treatment. Values below represent posttreatment performance minus pretreatment performance.
Time Frame: pretreatment= in the morning; postreatment= in the afternoon, 30 minutes after intranasal spray administration
Population: 30 subjects were analyzed. Subjects were randomized to either the experimental or placebo group.
Measure: Mean (Standard Deviation); unit: Words successfully recalled
Arm/Group | Placebo (1) | Single-Dose Intranasal Insulin
Number analyzed (Participants) | 15 | 15
Words successfully recalled | 4.9 (2.4) | 5.3 (3.5)

2. Primary Outcome: Improvement in Cognitive Function- HVLT-Delayed Recall (Number)
Description: Subjects performed the HVLT word recall task after a 20-minute delay before and after intranasal treatment. In the HVLT delayed recall task, participants were asked to recall the same list of 12 words dictated in the immediate recall task 20 minutes after the completion of the immediate recall task. Words successfully recalled after the 20-minute delay were measured. Values below represent posttreatment performance minus pretreatment performance.
Time Frame: pretreatment= in the morning; postreatment= in the afternoon, 30 minutes after intranasal spray administration
Population: 30 subjects were analyzed in this study. Subjects were randomized to either the experimental or placebo group.
Measure: Mean (Standard Deviation); unit: Words successfully recalled
Arm/Group | Placebo (1) | Single-Dose Intranasal Insulin
Number analyzed (Participants) | 15 | 15
Words successfully recalled | 1.1 (1.8) | 1.4 (1.7)

3. Primary Outcome: CPT d Score
Description: Subjects performed a computer-based test designed to measure sustained attention (attention to a specific stimuli over a period of several minutes) before and after intranasal treatment. During this test, participants respond as quickly as possible to any consecutive presentation of identical stimuli on the computer screen. The stimuli (2, 3, and 4-digit targets) were presented with increasing cognitive load in successive blocks. Correct responses, responses made to the second of 2 identical stimuli presented in a row, were scored as hits. False alarms were also recorded. The "d prime score" is a score given to each participant on a scale of 0.0- 1.0 in which discrimination sensitivity is measured. A score of zero equates to no sensitivity, whereas a score of 1.0 equates to perfect sensitivity. Values below represent postreatment performance minus pretreatment performance.
Time Frame: pretreatment= in the morning; postreatment= in the afternoon, 30 minutes after intranasal spray administration
Population: 30 subjects were analyzed. Subjects were randomized to either the experimental or placebo group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (1) | Single-Dose Intranasal Insulin
Number analyzed (Participants) | 15 | 15
units on a scale | 0.12 (0.55) | 0.29 (0.39)

4. Primary Outcome: Improvement in Cognitive Function- CPT Hits Rate (Proportion)
Description: Subjects performed a computer-based test designed to measure sustained attention before and after intranasal treatment. The task is described in the previous outcome measure ("CPT d score"). Hits rate refers to each participant's ability to correctly respond to two consecutive target presentations (i.e. correct responses). Hits rate was measured as a proportion of overall attempts (0= no hits, 1.0= 100% accuracy on hits). Values below represent posttreatment performance minus pretreatment performance.
Time Frame: pretreatment= in the morning; postreatment= in the afternoon, 30 minutes after intranasal spray administration
Population: 30 subjects were analyzed. Subjects were randomized either to the experimental or placebo group.
Measure: Mean (Standard Deviation); unit: Proportion of overall attempts
Arm/Group | Placebo (1) | Single-Dose Intranasal Insulin
Number analyzed (Participants) | 15 | 15
Proportion of overall attempts | 0.03 (0.15) | 0.09 (0.14)

5. Primary Outcome: Improvement in Cognitive Function- CPT Reaction Time of Hits (Milliseconds)
Description: Subjects performed a computer-based test designed to measure sustained attention before and after intranasal treatment. The task is described in detail in a previous outcome measure ("CPT d score"). Reaction time of hits refers to the average time each participant took to correctly respond to a stimuli in milliseconds. Values below represent posttreatment performance minus pretreatment performance.
Time Frame: pretreatment= in the morning; postreatment= in the afternoon, 30 minutes after intranasal spray administration
Population: 30 subjects were analyzed. Subjects were randomized to either the experimental or placebo group.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Placebo (1) | Single-Dose Intranasal Insulin
Number analyzed (Participants) | 15 | 15
Milliseconds | 8.5 (64.1) | -13.8 (82.9)

6. Primary Outcome: Improvement in Cognitive Function- CPT False Alarm Rate (Proportion)
Description: Subjects performed a computer-based test designed to measure sustained attention before and after intranasal treatment. The task is described in detail in a previous outcome measure ("CPT d score"). False alarm rate refers to the proportion of overall attempts that were characterized as incorrect responses (responses to two non-identical targets). Values below represent posttreatment performance minus pretreatment performance.
Time Frame: pretreatment= in the morning; postreatment= in the afternoon, 30 minutes after intranasal spray administration
Population: 30 subjects were analyzed. Subjects were randomized to either the experimental or placebo group.
Measure: Mean (Standard Deviation); unit: Proportion of overall attempts
Arm/Group | Placebo (1) | Single-Dose Intranasal Insulin
Number analyzed (Participants) | 15 | 15
Proportion of overall attempts | -0.03 (0.10) | 0.02 (0.05)

ADVERSE EVENTS:
Time Frame: 28 months
Arm/Group | Placebo (1) | Single-Dose Intranasal Insulin
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No